CLINICAL TRIAL: NCT00985894
Title: Comparison Between Asynchronous Online Care Model for the Management of Atopic Dermatitis With That of Face-to-Face, Office Visits
Brief Title: Comparison Between Asynchronous Online Care Model With Usual In Office Care for the Management of Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 200917162
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Atopic Dermatitis
Keywords: Teledermatology; Telemedicine; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teledermatology (Experimental): Online Telemedicine Group
  Interventions: Other: Online Teledermatology Care
- Usual Care (Active Comparator): Conventional in-office care
  Interventions: Other: Conventional in Office Care

INTERVENTIONS:
Other: Online Teledermatology Care — Patients randomized to the intervention group will have their scheduled follow-up visits online via store and forward teledermatology.
  Other Names: Health care service modality
  Arms: Teledermatology
Other: Conventional in Office Care — Patients randomized to the control group will have their scheduled follow-up visits via conventional in office care.
  Other Names: Health care service modality
  Arms: Usual Care

SUMMARY:
The purpose of this study is to determine if an asynchronous online model of teledermatology can achieve similar clinical outcomes as compared to conventional in-office care for the management of atopic dermatitis. The investigators also aim to determine the effects of this online care model on patient quality of life as well as patient and physician satisfaction.

The investigators' hypotheses include the following:

1. Compared to in-person visits, the online care model will result in similar clinical improvement in atopic dermatitis disease severity.
2. Compared to in-person visits, the online care model will result in similar improvements in quality of life.
3. Providers and subjects in the online group will achieve a similar level of overall satisfaction as those in the in-person group.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 4 years or older at time of consent, may be male or female.
* Meet the Hanifin diagnostic criteria for atopic dermatitis.
* Capable of giving informed consent (for patients less than 18 years of age, assent will be obtained from the minor and informed consent will be obtained from a legal guardian).
* Able to image their skin or have someone do it for them.
* Able to adhere to the study visit schedule and other protocol requirements.
* Have access to a computer with internet connection, a digital camera, and an e-mail address.

Exclusion Criteria:

* Non English speaking patients.
* Patients requiring systemic treatment (e.g., cyclosporine, phototherapy).
* Patients requiring close laboratory monitoring.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) | Every 8 weeks
Patient-oriented Eczema Measure (POEM) | Every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: April W Armstrong, MD, Principal Investigator — UC Davis Department of Dermatology
Locations (1):
- UC Davis Department of Dermatology, Sacramento, California, United States

REFERENCES:
- [Derived] Armstrong AW, Johnson MA, Lin S, Maverakis E, Fazel N, Liu FT. Patient-centered, direct-access online care for management of atopic dermatitis: a randomized clinical trial. JAMA Dermatol. 2015 Feb;151(2):154-60. doi: 10.1001/jamadermatol.2014.2299. PMID 25338198